CLINICAL TRIAL: NCT00703833
Title: A Double-Blind, Multicenter, Placebo-Controlled Study of MK0777 Gel Extrusion Module (GEM) 1.5 mg b.i.d. in the Treatment of Outpatients With Generalized Anxiety Disorder
Brief Title: A Study of MK0777 Gel Extrusion Module (GEM) in the Treatment of Outpatients With Generalized Anxiety Disorder (0777-019)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0777-019; MK0777-019; 2007_630
Record Dates: First submitted 2008-06-22; First posted 2008-06-24 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — 7-(1,1-dimethylethyl)-6-(2-ethyl-2H-1,2,4-triazol-3-ylmethoxy)-3-(2-fluorophenyl)-1,2,4-triazolo(4,3-b)pyridazine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Drug
  Interventions: Drug: MK0777
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo (unspecified)

INTERVENTIONS:
Drug: MK0777 — Days 1-3 3mg MK0777, Days 4-7 6 mg MK0777, Days 8-28 3, 6 or 9 mg MK0777
  Arms: 1
Drug: Placebo (unspecified) — matching placebo
  Arms: 2

SUMMARY:
The study will look at the effectiveness of MK0777 in patients with Generalized Anxiety Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Current diagnosis of Generalized Anxiety Disorder
* Age 18 - 70

Exclusion Criteria:

* Women who are pregnant, or breast-feeding
* Use of illicit drugs
* History of drug or alcohol dependence

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2002-09; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
Measure the reduction of anxiety | after 4 weeks and at end of study

SECONDARY OUTCOMES:
Safety and efficacy | throughout study and at end of study

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC